CLINICAL TRIAL: NCT05408611
Title: The Effect of Acupressure on Pain, Menstrual Symptoms, and General Comfort in Adolescents with Primary Dysmenorrhea: a Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Acupressure on Pain, Menstrual Symptoms, and General Comfort in Adolescents with Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ahu AKSOY, Research Assistant, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 000
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-10

CONDITIONS: Pain; Dysmenorrhea Primary; Signs and Symptoms
Keywords: Primary dysmenorrhea; acupressure; pain; menstrual symptoms; general comfort
MeSH Terms: conditions — Pain; Signs and Symptoms | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: Adolescents who agreed to participate in the study by signing the voluntary consent form after being informed about the study will be assigned to the study or placebo groups by matching the numbers on the envelope according to their school numbers. In the study, a researcher will determine the acupressure and placebo points to be applied in adolescents and this researcher will make the first cycle application. Therefore, the researcher cannot be blinded. However, the participants will practice and be blinded without knowing whether the points to be treated are the acupressure point or the placebo point. Thus, the research will be carried out as a single-blind randomized controlled trial. When the research is completed, the data of the control and study groups (coded as A or B) will be transferred to the computer environment by a researcher independent of the research, and the data will be analyzed by a statistician and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (acupressure) group (Experimental): Acupressure (complementary and integrative medicine method) Acupressure will be applied individually to the experimental group for 15 minutes three times a day for three menstrual cycles (approximately 3 months). Data collection forms will be applied 4 times in total, before the intervention, at the end of Cycle 1, cycle 2, and cycle 3 (each cycle is 28 days)
  Interventions: Other: Acupressure
- Plasebo group (Placebo Comparator): Placebo acupressure will be performed at any point within 1.5 cm of the actual acupressure points.
  Placebo acupressure will be applied individually to the placebo group for 15 minutes three times a day for three menstrual cycles (approximately 3 months). Data collection forms will be applied 4 times in total, before the intervention, at the end of Cycle 1, cycle 2, and cycle 3 (each cycle is 28 days)
  Interventions: Other: Placebo acupressure

INTERVENTIONS:
Other: Acupressure — acupressure is a non-pharmacological method originating from traditional Chinese medicine. According to the National Cancer Institute, acupressure is defined as pressure / massage applied to certain parts of the body to control symptoms such as pain or nausea. The main purpose of acupressure is to stimulate the regions associated with the specific organ by applying pressure with energy channels called meridians.
  Arms: Experimental (acupressure) group
Other: Placebo acupressure — Placebo acupressure is manual pressure applied to unreal acupressure points.
  Arms: Plasebo group

SUMMARY:
In this study, it is planned to determine the effect of acupressure applied to adolescents with primary dysmenorrhea on pain, menstrual symptoms and general comfort. The research questions of the research are as follows; Research Questions

* Is there a difference in pain scores in the post-acupressure intervention group and the placebo group?
* Is there a difference between menstrual symptoms scores in the post-acupressure intervention group and the placebo group?
* Is there a difference between comfort scores in the intervention group and the placebo group after acupressure?
* Is there a difference between the pain scores of the intervention group according to time?
* Is there a difference between the menstrual symptoms scores of the intervention group according to time?
* Is there a difference between the comfort scores of the intervention group according to time? Is there a difference between the pain scores of the placebo group over time? Is there a difference between the menstrual symptoms scores of the placebo group over time?
* Is there a difference between the comfort scores of the placebo group over time?

DETAILED DESCRIPTION:
Methods:

Adolescents aged 14-17 years with primary dysmenorrhea will be randomly assigned to the acupressure and control groups. The study group (n=26) and placebo group (n=26) will be applied to the determined points in a certain order. The order of application is Hegu (LI4), Zusanli (ST36), Sanyinjiao (SP6). Acupressure will be applied to the adolescents in the groups individually for 18-20 minutes, twice a day in the first three days of their menstrual periods. The primary outcome measures of the study is the effect of acupressure on adolescent pain severity and menstrual symptoms. The secondary outcome measures of the study is the effect of acupressure on general comfort. Data collection forms will be applied four times in total for the second and third cycles, before and immediately after the acupressure application.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 14-17,
* Willing to participate in the research,
* Open to communication,
* Having a regular menstrual period (occurring at intervals of 21-35 days and lasting 3-8 days),
* Menstrual pain severity is at least 4 according to the Visual Pain Scale,
* A score of 60 or more on the Menstruation Symptom Scale,
* Not using hormonal contraception and intrauterine device,
* Not pregnant and not experiencing pregnancy before,
* Does not have a systemic and chronic disease,
* Have not had a gynecological disorder or surgery before,
* Not using analgesics 6 hours before and during the study period,
* Body mass index <30 kg/m2
* No physical/mental health problems that would prevent/limit acupressure and exercise,
* Not doing regular acupressure,
* No psychiatric problems
* Adolescents without active COVID-19 infection.

Exclusion Criteria:

* Not between the ages of 14-17,
* Not willing to participate in the research,
* Closed to communication,
* Not having a regular menstrual period (not occurring at intervals of 21-35 days and lasting more or less than 3-8 days),
* Menstrual pain severity is less than 4 according to the Visual Pain Scale,
* A score below 60 on the Menstruation Symptom Scale,
* Using hormonal contraception and intrauterine device,
* Pregnant and experienced pregnancy before,
* Having a systemic and chronic disease,
* Have had a previous gynecological disorder or surgery,
* Using analgesics 6 hours before and during the study period,
* Body mass index ≥30 kg/m2
* Having physical/mental health problems that will prevent/limit acupressure and exercise,
* Regular acupressure
* Having a psychiatric problem
* Adolescents with active COVID-19 infection.

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | change from before the intervention, at the end of Cycle 1, cycle 2 and cycle 3 (each cycle is 28 days).
  Pain will be evaluated by using the "Visual Analog Skala (VAS)" . The Visual Analog Scale is used to measure the pain perceived by the person. There is a 10 cm mark on the one end of the scale, where there is no pain (zero), and on the other end there is the most severe (10) pain. Between the (100 mm.) part, the individual can indicate his or her pain by drawing a line, putting a dot or pointing. The distance from the point where there is no pain to the point marked by the individual is measured in centimeters, and the value found indicates the severity of the individual's pain. In the VAS scale, 0-44 mm indicates mild pain, 45-74 mm indicates moderate pain, while 75-100 mm indicates severe pain.
Menstrual Symptom Questionnaire (MSQ) | change from before the intervention, at the end of Cycle 1, cycle 2 and cycle 3 (each cycle is 28 days).
  Menstrual symptoms will be evaluated by using the "Menstrual Symptom Questionnaire ". The Menstrual Symptom Questionnaire was developed by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. The scale, which is a five-point Likert type and consists of 24 items, was updated by Negriff et al. in 2009 by re-evaluating its factor structure and usability. The MSQ score is calculated by taking the total mean score of the items in the scale. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The original Cronbach's Alpha value of the scale was .86 and had three sub-dimensions: "Negative Effects/Somatic Complaints", "Menstrual Pain" and "Abdominal Pain".
  The Turkish validity and reliability study of the Menstruation Symptom Questionnaire was performed by Güvenç et al. in 2014. Two items (6th and 17th items) in the original of the scale were removed from the scale because they had an item-total score correlation of less than 0.30. The scale

SECONDARY OUTCOMES:
General Comfort Scale (GAS) | change from before the intervention, at the end of Cycle 1, cycle 2 and cycle 3 (each cycle is 28 days).
  Comfort level will be evaluated by using the "General Comfort Scale (GAS)". It was developed by Kolcaba (1992) by taking the taxonomic structure, which includes three levels and four dimensions that make up the theoretical components of comfort, as a guide. The GAQ, which is suitable for Turkish society by Kuğuoğlu and Karabacak (2008), is of four and six-point Likert type, contains 24 positive and 24 negative items, and the response patterns are given in mixed form. The scale consists of three levels: relief (16 items), relaxation (17 items) and overcoming problems (15 items); It consists of four dimensions, namely the physical dimension (12 items), the psychospiritual dimension (13 items), the environmental dimension (13 items), and the sociocultural dimension (10 items). In the evaluation of the scale; Negative scores obtained are reverse coded and added up with positive items. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. The

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksoy-Can A, Buldum A, Abic A, Vefikulucay-Yilmaz D. The effect of acupressure on pain, menstrual symptoms, and comfort in adolescents with primary dysmenorrhea: a single-blind randomized controlled trial. BMC Complement Med Ther. 2025 Jul 2;25(1):221. doi: 10.1186/s12906-025-04965-0. PMID 40605053
- See also: The effects of acupressure on severity of primary dysmenorrhea — https://pmc.ncbi.nlm.nih.gov/articles/PMC3287417/
- See also: Effectıveness Of Abdomınal Stretchıng Exercıse And Sanyınjıao Acupressure To Relıeve Dysmenorrhea Paın — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5187401/